CLINICAL TRIAL: NCT00929526
Title: Long-term Extension Study of the Efficacy of the 580299 Vaccine in the Prevention of HPV-16 and/or HPV-18 Associated Cervical Intraepithelial Neoplasia (CIN) in Japanese Women Vaccinated in the Primary Vaccination Study NCT00316693
Brief Title: Extension Study of the Efficacy of the GSK 580299 Vaccine in Japanese Women Vaccinated in the Primary NCT00316693 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112949
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine; cervical intraepithelial neoplasia (CIN); including new onset of autoimmune disease [NOAD]); new onset of chronic disease (NOCD); medically significant condition (MSC)
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia | interventions — AKAP13 protein, human; Blood Specimen Collection

ARMS (2):
- Cervarix Group (Experimental): subjects received 3 doses of Cervarix™ vaccine in primary vaccination study NCT00316693.
  Interventions: Procedure: Liquid-based cytology (LBC) sampling; Procedure: Blood sampling
- Aimmugen Group (Placebo Comparator): subjects received 3 doses of Aimmugen ™ vaccine in primary vaccination study NCT00316693.
  Interventions: Procedure: Liquid-based cytology (LBC) sampling

INTERVENTIONS:
Procedure: Liquid-based cytology (LBC) sampling — LBC samples will be collected at Months 36 and 48 for cytology and HPV DNA testing (by PCR)
Procedure: Blood sampling — Blood samples will be collected at Months 36 and 48 for antibody determination
  Arms: Cervarix Group

SUMMARY:
This extension study is conducted to assess the efficacy of the GSK 580299 vaccine against cervical intraepithelial neoplasia (CIN) lesions, cervical cancer and cytological abnormalities associated with human papillomavirus (HPV)-16 and/or HPV-18 or other oncogenic HPV types for an additional two years. All subjects who participated in the primary vaccination study NCT00316693 and who confirmed their interest in participating in a long term follow up study will therefore be invited to be followed for up to 48 months after administration of the first dose of vaccine. In addition, safety and persistence of the humoral immune response will be evaluated in this study.

This protocol posting deals with objectives & outcome measures of the extension phase at Months 36 and 48. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00316693).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol;
* Written informed consent obtained from the subject prior to enrolment in the extension study;
* A subject previously vaccinated in the NCT00316693 study.
* Subjects who showed, at the last NCT00316693 study visit (at Month 24) willingness to participate in this extension study.

Exclusion Criteria:

* Use of any HPV vaccine other than the one administered in the NCT00316693 study;
* Use of any investigational or non-registered product other than the study vaccine since last NCT00316693 study visit, or planned use during the study period;
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product;
* Subjects who were diagnosed high grade or missing cytology at Month 0 in the NCT00316693 study;
* Pregnant females and females who were pregnant less than 3 months ago.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 752 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Japan (7):
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chen J, Gopala K, Akarsh PK, Struyf F, Rosillon D. Prevalence and Incidence of Human Papillomavirus (HPV) Infection Before and After Pregnancy: Pooled Analysis of the Control Arms of Efficacy Trials of HPV-16/18 AS04-Adjuvanted Vaccine. Open Forum Infect Dis. 2019 Dec 4;6(12):ofz486. doi: 10.1093/ofid/ofz486. eCollection 2019 Dec. PMID 31824976
- [Derived] Konno R, Yoshikawa H, Okutani M, Quint W, V Suryakiran P, Lin L, Struyf F. Efficacy of the human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical intraepithelial neoplasia and cervical infection in young Japanese women. Hum Vaccin Immunother. 2014;10(7):1781-94. doi: 10.4161/hv.28712. PMID 25424783
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112949 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No vaccines were administered in this extension study. The mean duration of this study was aproximately 12 months for each subjects (from Month 0 up to Month 12). This study began 36 months after the first vaccination in study NCT00316693.
Pre-assignment Details: Subjects were randomised in the primary vaccination study NCT00316693 to receive the Cervarix vaccine or the Aimmugen vaccine and were aged 20 - 25 years at the time of first vaccination. Only subjects showing willingness to participate in this long term follow-up study and who had signed the informed consent form entered this study.
Period: Overall Study
Arm/Group | Cervarix Group | Aimmugen Group
Started | 375 | 377
Completed | 358 | 348
Not Completed | 17 | 29
Not completed — Withdrawal by Subject | 1 | 11
Not completed — Lost to Follow-up | 8 | 12
Not completed — Other | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Aimmugen Group | Total
Number analyzed (Participants) | 375 | 377 | 752
Age, Continuous [Mean (Standard Deviation); unit: Years] — Japanase women aged 20 to 25 years at the time of first vaccination in the primary study NCT00316693
  Years | 25.4 (1.72) | 25.5 (1.72) | 25.5 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 377 | 752
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Cases Associated With HPV16 and/or HPV18 Detected Within the Lesional Component of the Cervical Tissue Specimen.
Description: Low-grade cervical lesions and higher lesions are defined as CIN1+, i.e. CIN grade 1 (CIN1), CIN grade 2 (CIN2), CIN grade 3 (CIN3), adenocarcinoma in situ (AIS) or invasive cervical cancer (ICC).
  Detection of vaccine oncogenic Human papillomavirus (HPV) types 16 or 18 was made by polymerase chain reaction (PCR).
  For single type: Subjects Deoxyribonucleic acid (DNA) negative at Month 0 and Month 6 and seronegative at Month 0 for the corresponding HPV type.
  For combined types: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for at least one HPV type.
Time Frame: From Month 0 up to Month 12
Population: The analysis was performed in subjects who were seronegative at baseline and negative for human papillomavirus (HPV) desoxyribonucleic acid (DNA) at baseline and Month 6 in the primary study (NCT00316693) for the HPV-type considered and for whom data concerning efficacy outcome measures were available in this follow-up study.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 332 | 335
Subjects
  CIN1+ HPV-16/18 (N=332;335) | 0 | 5
  CIN1+ HPV-16 (N=286;289) | 0 | 5
  CIN1+ HPV-18 (N=294;291) | 0 | 0

2. Secondary Outcome: Number of Subjects Reporting Cytological Abnormalities and Lesions Associated With HPV-16 and/or HPV-18.
Description: Cytologically confirmed abnormalities and lesions (ASC-US+) are defined as atypical squamous cell of undetermined significance (ASC-US), low-grade squamous intraepithelial lesions (LSIL), high-grade squamous intraepithelial lesions (HSIL), atypical squamous cell-cannot exclude HSIL (ASC-H) and atypical glandular cells (AGC).
  For single type: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for the corresponding HPV type.
  For combined types: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for at least one HPV type.
Time Frame: From Month 0 up to Month 12
Population: The analysis was performed in subjects who were seronegative at baseline and negative for HPV DNA at baseline and Month 6 in the primary study (NCT00316693) for the HPV-type considered and for whom data concerning efficacy outcome measures were available in this follow-up study.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 332 | 335
Subjects
  ASC-US+ HPV-16/18 (N=332;335) | 3 | 11
  ASC-US+ HPV-16 (N=286;289) | 2 | 10
  ASC-US+ HPV-18 (N=294;291) | 1 | 2

3. Secondary Outcome: Number of Subjects Reporting Cytologically Confirmed Abnormalities and Lesions Concurrently Associated With Any Oncogenic HPV Types.
Description: Cytologically confirmed abnormalities and lesions (ASC-US+) are defined as ASC-US, LSIL, HSIL, ASC-H and AGC.
  HR= High-risk HPV-types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: From Month 0 up to Month 12
Population: The analysis was performed in subjects who were DNA negative at baseline and Month 6 in the primary study (NCT00316693) for the HPV-type considered, regardless of their initial serostatus and for whom data concerning efficacy outcome measures were available in this current follow-up study.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 363 | 359
Subjects | 33 | 45

4. Secondary Outcome: Number of Subjects Reporting CIN1+ Associated With Any Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen.
Description: Low-grade cervical lesions and higher lesions are defined as CIN1+, i.e. CIN1, CIN2, CIN3, AIS or ICC.
  HR=High-risk HPV-types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: From Month 0 up to Month 12
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 363 | 359
Subjects | 8 | 22

5. Secondary Outcome: Number of Subjects Reporting Incident Cervical Infection Associated With HPV-16 and/or 18.
Description: For single type: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for the corresponding HPV type.
  For combined types: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for at least one HPV type.
Time Frame: From Month 0 up to Month 12
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 332 | 335
Subjects
  Incident infection HPV-16/18 (N=332;335) | 7 | 28
  Incident infection HPV-16 (N=286;289) | 3 | 16
  Incident infection HPV-18 (N=294;291) | 5 | 13

6. Secondary Outcome: Number of Subjects Reporting Incident Cervical Infection With Any Oncogenic HPV Types.
Description: HR=High-risk HPV-types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: From Month 0 up to Month 12
Population: The analysis was performed in subjects who were negative for HPV DNA at baseline and Month 6 in the primary study (NCT00316693) for the HPV-type considered, regardless of their initial serostatus and for whom data concerning efficacy outcome measures were available in this current follow-up study.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 363 | 359
Subjects | 87 | 98

7. Secondary Outcome: Number of Subjects Reporting Persistent Long-term Cervical Infection (12-month Definition) With HPV-16 and/or 18.
Description: Persistent infection (12-month definition): detection of at least 2 positive HPV DNA PCR assays for the same viral genotype with no negative DNA sample between the 2 positive DNA samples, over an approximate interval of 12 months (>300 days).
  For single type: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for the corresponding HPV type.
  For combined types: Subjects DNA negative at Month 0 and Month 6 and seronegative at Month 0 for at least one HPV type.
Time Frame: From Month 0 up to Month 12
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 257 | 241
Subjects
  Persistent infection HPV-16/18 (N=257;241) | 0 | 9
  Persistent infection HPV-16 (N=225;206) | 0 | 6
  Persistent infection HPV-18 (N=227;209) | 0 | 4

8. Secondary Outcome: Number of Subjects Reporting Persistent Long-term Cervical Infection (12-month Definition) With Any Oncogenic HPV-types.
Description: Persistent infection: subjects with at least 2 positive samples (difference > than 300 days) and no negative samples in between.
  HR=High-risk HPV-types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: From Month 0 up to Month 12
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 280 | 261
Subjects | 19 | 31

9. Secondary Outcome: Number of Subjects With HPV-16 and HPV-18 Antibodies Titers Equal to or Above the Assay Cut-off Values.
Description: Assay cut-off values assessed were 8 Enzyme-linked Immunosorbent Assay (ELISA) units per millilitre (EL.U/mL) for HPV-16 antibodies and 7 ELISA units per millilitre (EL.U/mL) for HPV-18 antibodies in the Cervarix Group.
Time Frame: At Month 0 and at Month 12
Population: The According-To-Protocol cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome measures were available in this current follow-up study for antibodies against at least one study vaccine antigen component.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 291 | 0
Subjects
  HPV-16 >=8 EL.U/mL [at Month 0] (N=282) | 282 |
  HPV-16 >=8 EL.U/mL [at Month 12] (N=291) | 291 |
  HPV-18 >=7 EL.U/mL [at Month 0] (N=281) | 281 |
  HPV-18 >=7 EL.U/mL [at Month 12] (N=290) | 290 |

10. Secondary Outcome: HPV-16 and HPV-18 Antibody Titers
Description: Titers were expressed as Geometric Mean Titers (GMTs). Geometric mean titres were assessed by ELISA in the Cervarix Group.
Time Frame: At Month 0 and at Month 12
Population: The According-To-Protocol cohort for immunogenicity M48 EXT- NCT00316693 included all evaluable subjects for whom data concerning immunogenicity outcome measures were available in this current follow-up study for antibodies against at least one study vaccine antigen component.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 291 | 0
Titers
  HPV-16 [Month 0] (N=282) | 1409.9 [1268.1 to 1567.6] |
  HPV-16 [Month 12] (N=291) | 1294.8 [1171.4 to 1431.1] |
  HPV-18 [Month 0] (N=281) | 572.3 [505.6 to 647.7] |
  HPV-18 [Month 12] (N=290) | 470.9 [419.2 to 528.9] |

11. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the follow-up period from last study visit at Month 24 in the primary vaccination study NCT00316693 until the end of this follow-up study at Month 12
Population: The analysis was performed on all subjects from the Total Vaccinated cohort who came for the current follow-up study and for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 375 | 377
Subjects | 11 | 16

12. Secondary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs) Regardless of Causal Relationship to Vaccination and Intensity.
Description: NOCDs included autoimmune diseases, diabetes mellitus.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 375 | 377
Subjects | 2 | 2

13. Secondary Outcome: Number of Subjects With New Onset of Autoimmune Diseases (NOADs) Regardless of Causal Relationship to Vaccination and Intensity.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 375 | 377
Subjects | 2 | 1

14. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSCs).
Description: MSCs were defined as adverse events (AEs) prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that were not related to common disease.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 375 | 377
Subjects | 11 | 15

15. Secondary Outcome: Number of Subjects With Pregnancies and Pregnancy Outcomes.
Description: Pregnancy outcomes are live infant, elective termination, ectopic pregnancy, stillbirth, spontaneous abortion, lost to follow-up and pregnancy ongoing. For each category it was specified if the infant presents congenital anomaly (CA) or no apparent congenital anomaly (No ACA).
Time Frame: During the follow-up period from last study visit at Month 24 in the primary vaccination study NCT00316693 until the end of this follow-up study at Month 12 (Month 48 Ext- NCT00316693).
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Aimmugen Group
Number analyzed (Participants) | 37 | 41
Subjects
  Live infant No ACA | 28 | 30
  Live infant CA | 0 | 1
  Elective termination No ACA | 4 | 3
  Spontaneous abortion No ACA | 3 | 4
  Stillbirth No ACA | 1 | 0
  Ectopic pregnancy | 0 | 1
  Lost to follow-up | 0 | 2
  Pregnancy ongoing | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs: from Month 24 (last study visit in the primary vaccination study NCT00316693) until Month 12 in this current follow-up study.
Description: The analysis was performed on all subjects from the Total Vaccinated cohort who came for the current follow-up study and for whom data were available. Other adverse events (solicited and unsolicited) were not assessed and not reported during this study.
Arm/Group | Cervarix Group | Aimmugen Group
Serious Adverse Events (participants affected / at risk) | 11/375 | 16/377
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=375) | Aimmugen Group (N=377)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Allergic granulomatous angiitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 0 | 1
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.